CLINICAL TRIAL: NCT02504125
Title: The Efficacy and Safety of Using Tranexamic Acid to Reduce Blood Loss In Simultaneous Bilateral Total Knee Arthroplasty: a Randomized, Double-blind, Controlled Trial
Brief Title: The Efficacy and Safety of Using Tranexamic Acid to Reduce Blood Loss In Simultaneous Bilateral Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chenxiaoyong, Doctor-in-charge, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJODCT2014002
Record Dates: First submitted 2015-06-23; First posted 2015-07-21 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Receving TXA, Study group (Experimental): Tranexamic acid, Study group tranexamic acid 1g, intravenous injection, pre-operationally
  Interventions: Drug: Tranexamic Acid
- Normal saline, Control group (Placebo Comparator): Not receiving tranexamic acid, Control group Normal saline 100mL, intravenous injection, pre-operationally
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid — 1 g of tranexamic acid in 100 mL of normal saline intravenously approximately 15 minutes before incision
  Arms: Receving TXA, Study group
Drug: Normal saline — 100 mL of normal saline intravenously approximately 15 minutes before incision
  Arms: Normal saline, Control group

SUMMARY:
A randomized, double-blind, single-center and controlled study comparing the efficacy and safety of intravenous administration of tranexamic acid to reduce blood loss in simultaneous bilateral total knee arthroplasty.

DETAILED DESCRIPTION:
A randomized, double-blind, single-center and controlled study comparing the efficacy and safety of intravenous administration of tranexamic acid to reduce blood loss in simultaneous bilateral total knee arthroplasty. Subjects will be monitored for occurrence of any complications, particularly deep venous thrombosis and thromboembolism during the hospital stay and for 1 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who plan to undergo simultaneous primary total knee arthroplasty on bilateral knee joint with a diagnosis of osteoarthritis or aseptic bone necrosis, but not of rheumatoid arthritis;
* All patients who have normal preoperative platelet count, normal prothrombin time, normal partial thromboplastin time, and normal international normalized ratio;
* The use of only balanced electrolyte solutions and/or albumin for plasma volume restitution

Exclusion Criteria:

* Allergy to tranexamic acid;
* Receiving warfarin or heparin; had a history of hemophilia, deep venous thrombosis, pulmonary embolism, or renal impairment; or were pregnant;
* Patients with any cardiovascular problems (such as myocardiac infarction history, atrial fibrillation, angina);
* Patients with thromboembolic disorders, or those exhibiting a deteriorating general condition;
* Preoperative anemia (a hemoglobin value of <11 g/dL in females and <12 g/dL in males), refusal of blood products;
* Preoperative use of anticoagulant therapy within five days before surgery, fibrinolytic disorders requiring intraoperative antifibrinolytic treatment, coagulopathy (as identified by a preoperative platelet count of <150,000/mm3, an international normalized ratio of >1.4, or a prolonged partial thromboplastin time [>1.4 times normal]).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rate of Allogeneic Blood Transfusion as a Measure of Efficacy | one week after surgery

SECONDARY OUTCOMES:
Amount of Total Blood Loss as a Measure of Efficacy | one week after surgery
Rate of Thrombotic Complications as a Measure of Safety | 1 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Zhu, M.D., Study Director — Department of Orthropaedics, Xijing Hospital
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China